CLINICAL TRIAL: NCT06394921
Title: Interrogative Approaches Identify Causes of Physical Impairment in Those Affected by Post COVID-19 Morbidity (Long COVID) - an International Multicenter Observational Study
Brief Title: Cardiopulmonary Exercise Tests in Patients With Long COVID
Acronym: PREPP-19
Status: Completed | Type: Observational
Sponsor: Sheffield Hallam University (Other)
Collaborators: MS Ramaiah Medical College & Hospitals (Other); University of Illinois at Chicago (Other); University of Nottingham (Other); Northumbria University (Other); King's College London (Other); University of Derby (Other)
Responsible Party: Sponsor
Other Study IDs: PREPP19
Record Dates: First submitted 2024-03-26; First posted 2024-05-01 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Long COVID; COVID Long-Haul
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with Long COVID: Eligibility
  * Aged 18 to 65 years old
  * Diagnosed with COVID-19
  * Still suffering from symptoms and experiencing functional limitations beyond 3 months after initial COVID-19 infection (quantified as PCFS grade 1 or greater).
  * Sufficient English language comprehension and cognitive ability to understand the study protocol, give informed consent and follow instructions.
  Interventions: Procedure: 2 day cardiopulmonary exercise test

INTERVENTIONS:
Procedure: 2 day cardiopulmonary exercise test — Consecutive day 2 day CPET and follow up for 7 days for subjective feelings/fatigue.

SUMMARY:
The value of clinical cardiopulmonary exercise testing (CPET) within healthcare settings has been established in the last decade. CPET methods remain highly relevant in the COVID-19 endemic phase and should be used to assess those recovering from COVID-19 (SARS-CoV-2) infection. This diagnostic tool could play an integral role in disease prognostication and evaluate the integrative response to incremental exercise. Date from such assessments can enable practitioners to characterise cardio-respiratory fitness and identify reasons for physical impairment or abnormal cardio-respiratory function. More than 50% of patients admitted to hospital will experience cardiorespiratory issues and significant morbidity during their recovery and will require significant rehabilitative support. In this context, measurements obtained from an assessment of cardio-respiratory responses to physiological stress could provide insight regarding the integrity of the pulmonary-vascular interface and characterisation of any impairment or abnormal cardio-respiratory function. Current approaches to rehabilitation are being developed on existing knowledge from Severe Acute Respiratory Syndrome (SARS) and Acute Respiratory Distress Syndrome (ARDS) related illness. These provide important insight but do not provide insight into the novel challenges provided by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* • Aged 18 to 65 years old

  * Diagnosed with COVID-19
  * Still suffering from symptoms of COVID-19, 3 months after initial infection
  * Sufficient English language comprehension and cognitive ability to understand the study protocol, give informed consent and follow instructions.

Exclusion Criteria:

* • <18 years of age

  * Admitted to or received treatment from Intensive Care Units
  * Unconfirmed COVID-19 test diagnosis
  * Unable to understand verbal or written information in English
  * Achieving a grade 0 or 1 on the PCFS.
  * Unstable angina
  * Uncontrolled hypertension, that is, resting systolic blood pressure (SBP) >180mmHg, or resting diastolic blood pressure (BP) (DBP) >110mmHg
  * Orthostatic blood pressure drop of >20 mmHg with symptoms
  * Significant aortic stenosis (aortic valve area 120 bpm)
  * Acute pericarditis or myocarditis
  * Decompensated HF
  * Third degree (complete) atrioventricular (AV) block without pacemaker
  * Recent embolism
  * Acute thrombophlebitis
  * Resting ST segment displacement (>2 mm)
  * Uncontrolled diabetes mellitus
  * Severe orthopaedic conditions that would prohibit exercise
  * Other metabolic conditions, such as acute thyroiditis, hypokalaemia, hyperkalaemia or hypovolaemia (until adequately treated)
  * Severe grade 3 rejection (cardiac transplantation recipients Appendix N).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be assessed according to the eligibility criteria and recruited directly from Long COVID Clinics in the UK (Derbyshire Community Health Services, Sheffield Teaching Hospitals NHS Foundation Trust and Northumbria NHS Trust), the University of Illinois Post-COVID-19 Clinic, (Chicago, USA) and the Ramiah Medical Centre Post COVID Centre (Bangalore, India). Long COVID patients will be assessed according to the eligibility criteria and recruited following referral or contact with a long COVID clinic or having suspected or confirmed long COVID. Social media and targeted recruitment from established pages will be used to advertise the opportunity to engage with the trial for those in proximity
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Test- Rate of Oxygen Utilisation | During CPET1 and CPET2
  Rate of Oxygen Utilisation (VO2; l/min)
Cardiopulmonary Exercise Test- Rate of carbon dioxide production | During CPET1 and CPET2
  Rate of Carbon Dioxide Production (VCO2; l/min)
Cardiopulmonary Exercise Test- Respiratory Exchange Ratio | During CPET1 and CPET2
  Respiratory Exchange Ratio (VO2/VCO2)
Cardiopulmonary Exercise Test: Maximal Rate of Oxygen Utilisation | During CPET1 and CPET2
  Maximal Rate of Oxygen Utilisation per kg body mass (VO2max; ml/kg/min)
Cardiopulmonary Exercise Test- Respiratory Threshold | During CPET1 and CPET2
  Respiratory Threshold breath by breath (l/min)
Cardiopulmonary Exercise Test- Minute Ventilation | During CPET1 and CPET2
  Minute Ventilation using breath by breath (l/min)
Cardiopulmonary Exercise Test- Blood lactate | During CPET1 and CPET2
  Blood Lactate Concentration from fingertip (mmol/l)
Prevalence of symptoms of post exertional Malaise | 7 days post exercise
  Symptom Profile post exercise protocols- Questionnaire

SECONDARY OUTCOMES:
Blood biomarkers of Inflammation- IL-6 | Day 1 and Day 2
  Concentration of Interleukin 6
Blood biomarkers of Inflammation- IL-1 | Day 1 and Day 2
  Concentration of Interleukin 1
Blood biomarkers of Inflammation- Microclots | Day 1 and Day 2
  Number of Microclots
Blood biomarkers of Inflammation- D-Dimer | Day 1 and Day 2
  D-Dimer Concentration
Blood biomarkers of Inflammation- CRP | Day 1 and Day 2
  C-Reactive protein Concentration
Echocardiogram | Baseline, Day 1 and Day 2
  12 lead echocardiogram.
Resting Systolic Blood Pressure | Baseline, Day 1 and Day 2
  Systolic Blood Pressure at Rest (mmHg)
Resting Diastolic Blood Pressure | Baseline, Day 1 and Day 2
  Diastolic Blood Pressure at Rest (mmHg)
Exercise Diastolic Blood Pressure | Baseline, Day 1 and Day 2
  Diastolic Blood Pressure During Exercise (mmHg)
Exercise Systolic Blood Pressure | Baseline, Day 1 and Day 2
  Systolic Blood Pressure During Exercise (mmHg)

OTHER OUTCOMES:
Symptom Profile Questionnaire | Baseline
  Description of previous and current symptom/s of Long COVID
Quality of Life questionnaire | Baseline
  EQ-5D-5L
Sleep Behavour | Baseline
  Pittsburgh Sleep Quality Index
Fatigue Questionnaire- FAS | Baseline, Day 1 and Day 2
  Fatigue Assessment Scale
Fatigue Questionnaire- MFI | Baseline, Day 1 and Day 2
  Multidimensional Fatigue Index (MFI-20)
Medical Research Council Dyspnoea Scale | Baseline
  Breathlessness scale
Post COVID-19 functional status Scale | Baseline
  Questionnaire to see effect of COVID-19 on physical function- 0= No Limitations; 4- Severe Limitations to function
Cognition | Baseline
  Montreal cognitive assessment
6 minute walk | Baseline
  6 minute walk distance (metres)
Timed Up and Go | Baseline
  5m timed up and go (seconds)
Lung Function Assessment- FEV1 | Baseline
  Forced Expiratory Volume in 1 Second (l)
Lung Function Assessment- FVC | Baseline
  Forced Vital Capacity (l)
Lung Function Assessment- PEF | Baseline
  Peak Expiratory Flow Rate (l/min)
Lung Function Assessment- MIP | Baseline
  Maximal Inspiratory Pressure (mmHg)
Lung Function Assessment- MEP | Baseline
  Maximal Expiratory Pressure (mmHg)
Height | Baseline
  measurement of body stature (m)
Weight | Baseline
  Measurement of body mass (kg)
body mass index | Baseline
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (5):
- University of Illinois at Chicago, Chicago, Illinois, United States
- Ramaiah Medical College, Bengaluru, India
- United Kingdom (3):
  - University of Derby, Derby, Derbyshire
  - Sheffield Hallam University, Sheffield, South Yorkshire
  - Northumbria University, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT06394921/Prot_000.pdf